CLINICAL TRIAL: NCT00268892
Title: An Open-Label, Multi-Centre, Extension Study, Evaluating the Long-Term Safety and Tolerability of Different Three-Month Degarelix Dosing Regimens in Patients With Prostate Cancer
Brief Title: Extension Study Investigating the Long-Term Safety of Degarelix Three-Month Depots in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS15A
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Results first posted 2010-12-06 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen ablation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Degarelix 240/240@40(1-3-6-9) (Experimental): Participants in this arm who completed the main study continued with the same dose (240 mg (40 mg/mL) starting dose and 240 mg (40 mg/mL) at months 1, 3, 6, and 9) in the extension study (240 mg (40 mg/mL) every three months). A protocol amendment in June 2006 changed the dosage to 360 mg or 480 mg (60 mg/mL).
  Interventions: Drug: Degarelix
- Degarelix 240/240@60(1-3-6-9) (Experimental): Participants in this arm who completed the main study continued with the same dose (240 mg (40 mg/mL) starting dose and 240 mg (60 mg/mL) at months 1, 3, 6, and 9) in the extension study (240 mg (60 mg/mL) every three months). A protocol amendment in June 2006 changed the dosage to 360 mg or 480 mg (60 mg/mL).
  Interventions: Drug: Degarelix
- Degarelix 240/240@60(1-4-7-10) (Experimental): Participants in this arm who completed the main study continued with the same dose (240 mg (40 mg/mL) starting dose and 240 mg (60 mg/mL) at months 1, 4, 7, 10) in the extension study (240 mg (60 mg/mL) every three months). A protocol amendment in June 2006 changed the dosage to 360 mg or 480 mg (60 mg/mL).
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Participants who completed the main study initially continued with the same dose in the FE200486 CS15A extension study. A protocol amendment changed the dosage to 360 mg (60 mg/mL) or 480 mg (60 mg/mL).
  Drug supplied as a powder to be dissolved in the solvent for solution for injection. Degarelix given by subcutaneous injection every 3 months until the end of the study.
  Other Names: FE200486
  Arms: Degarelix 240/240@40(1-3-6-9)
Drug: Degarelix — Participants who completed the main study initially continued with the same dose in the FE200486 CS15A extension study. A protocol amendment changed the dosage to 360 mg (60 mg/mL) or 480 mg (60 mg/mL).
  Drug supplied as a powder to be dissolved in the solvent for solution for injection. Degarelix given by subcutaneous injection every 3 months until the end of the study.
  Other Names: FE200486
  Arms: Degarelix 240/240@60(1-3-6-9)
Drug: Degarelix — Participants who completed the main study initially continued with the same dose in the FE200486 CS15A extension study. A protocol amendment changed the dosage to 360 mg (60 mg/mL) or 480 mg (60 mg/mL).
  Drug supplied as a powder to be dissolved in the solvent for solution for injection. Degarelix given by subcutaneous injection every 3 months until the end of the study.
  Other Names: FE200486
  Arms: Degarelix 240/240@60(1-4-7-10)

SUMMARY:
The purpose of this extension study was to collect long-term safety and tolerability information to support a marketing authorisation application for a three-month dosage regimen of degarelix.

DETAILED DESCRIPTION:
The data include data from the participants who participated in both the main study FE200486 CS15 (NCT00113753) and the extension study FE200486 CS15A.

ELIGIBILITY:
Inclusion Criteria:

* Has given written consent prior to any study-related activity is performed. A study-related activity is defined as any procedure that would not have been performed during the normal management of the patient.
* Has successfully completed the main study.

Exclusion Criterion:

- Has been withdrawn from the main study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (23):
- UZ Gasthuisberg Leuven, Leuven, Belgium
- Finland (4):
  - Helsinki University Hospital, Maria Hospital, Building 11, Helsinki
  - Central Hospital, North Karelian, Joensuu
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
- Fédération d'Urologie et Néphrologie, BP69 Hôpital Pasteur, Nice, France
- Gemeinschaftspraxis Dres Effert und Benedic, Aachen, Germany
- Clinical Center Novi Sad, Clinic of Urology, Novi Sad, Montenegro
- Netherlands (2):
  - Academic Medical Center, Urology, Amsterdam
  - St. Elisabeth Hospital, Tilburg
- Romania (3):
  - "Centrul Medical Privat" Prof. Dr. Ioiart Ioan", Arad
  - Clinical Hospital "Prof. Dr. Theodor Burghele", Urology Department, Bucharest
  - University CF Hospital No. 2, Bucharest
- Russia (5):
  - Andros Clinic, Saint Petersburg
  - City Hospital #15, Saint Petersburg
  - City Hospital #26, Saint Petersburg
  - Pavlov State Medical University, Outpatient Diagnostic Center affiliated with the Urology Department, Saint Petersburg
  - Pavlov State Medical University, Urology Department, Saint Petersburg
- Clinical Center of Serbia, Institute of Urology and Nephrology, Belgrade, Serbia
- United Kingdom (4):
  - Mount Vernon Cancer Centre, Marie Cuire Research Wing, Northwood, Middlesex
  - Castle Hill Hospital, Hull, North Humberside
  - Ward 13, NHS Forth Valley Acute Operating Division, Falkirk and District Royal Infirmary, Majors Loans, Falkirk
  - Level 7, Urology Research Unit, Derriford Hospital, Plymouth

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the main FE200486 CS15(NCT00113753) study (except those in US and Canada) were asked to continue into the FE200486 CS15A extension study.
Pre-assignment Details: 447 participants started and 374 participants completed the main CS15 study. Of these, 278 participants were recruited into the extension study CS15A and 203 participants signed the informed consent for dose shift.
Period: Overall Study
Arm/Group | Degarelix 240/240@40(1-3-6-9) | Degarelix 240/240@60(1-3-6-9) | Degarelix 240/240@60(1-4-7-10)
Started | 90 | 95 | 93
Switched to Higher Dose | 59 | 68 | 76
Completed | 51 | 53 | 54
Not Completed | 39 | 42 | 39
Not completed — Adverse Event | 14 | 17 | 20
Not completed — Lack of Efficacy | 1 | 3 | 0
Not completed — Withdrawal by Subject | 14 | 15 | 13
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Lost to Follow-up | 5 | 2 | 4
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Disease Progression | 1 | 1 | 0
Not completed — Trial Site Closed | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 240/240@40(1-3-6-9) | Degarelix 240/240@60(1-3-6-9) | Degarelix 240/240@60(1-4-7-10) | Total
Number analyzed (Participants) | 90 | 95 | 93 | 278
Age Continuous [Mean (Standard Deviation); unit: years] — Safety analysis set.
  years | 72.7 (6.55) | 73.3 (7.00) | 71.8 (7.05) | 72.6 (6.88)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety analysis set.
  Participants
    Female | 0 | 0 | 0 | 0
    Male | 90 | 95 | 93 | 278
Race (NIH/OMB) [Count of Participants; unit: Participants] — Safety analysis set.
  Participants
    American Indian or Alaska Native | 0 | 0 | 1 | 1
    Asian | 0 | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 3 | 5 | 3 | 11
    White | 87 | 89 | 88 | 264
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: kilogram] — Safety analysis set.
  kilogram | 76.7 (13.0) | 76.9 (12.2) | 76.5 (12.8) | 76.7 (12.6)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] — Safety analysis set.
  kilogram per square meter | 25.4 (4.14) | 25.8 (3.93) | 25.8 (4.16) | 25.7 (4.07)
Curative Intent [Number; unit: participants] — Safety analysis set. A curative intent of Yes refers to participants who have been castrated via radical prostatectomy or radiotherapy.
  participants
    Yes | 10 | 12 | 7 | 29
    No | 80 | 83 | 86 | 249
Gleason Score [Number; unit: participants] — Safety analysis set. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive. A Gleason Score was missing for one participant in the Degarelix 240/240@60(1-3-6-9) group.
  participants
    2-4 | 13 | 6 | 13 | 32
    5-6 | 33 | 30 | 34 | 97
    7-10 | 44 | 58 | 46 | 148
Stage of Prostate Cancer [Number; unit: participants] — Safety analysis set. Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localized | 34 | 37 | 36 | 107
    Locally Advanced | 26 | 26 | 28 | 80
    Metastatic | 16 | 19 | 20 | 55
    Not Classifiable | 14 | 13 | 9 | 36
Time since Prostate Cancer Diagnosis [Mean (Standard Deviation); unit: days] — Safety analysis set.
  days | 469 (1079) | 347 (824) | 255 (583) | 356 (852)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Markedly Abnormal Values in Vital Signs and Body Weight
Description: This outcome measure included incidence of markedly abnormal values in blood pressure (systolic and diastolic), pulse, and body weight during the trial. The table presents the number of participants with a normal baseline value and at least one post-baseline markedly abnormal value.
Time Frame: Baseline and up to 4.5 years
Population: The data include data from participants participating in both the main study (FE200486 CS15) and the extension study FE200486 CS15A.
Measure: Number; unit: participants
Arm/Group | Degarelix 240/240@40(1-3-6-9) | Degarelix 240/240@60(1-3-6-9) | Degarelix 240/240@60(1-4-7-10)
Number analyzed (Participants) | 90 | 95 | 93
participants
  Diastolic blood pressure <=50 and decrease >=15 | 5 | 6 | 4
  Diastolic blood pressure >=105 and increase >=15 | 7 | 6 | 8
  Systolic blood pressure <=90 and decrease >=20 | 1 | 1 | 2
  Systolic blood pressure >=180 and increase >=20 | 8 | 11 | 10
  Heart rate <=50 and decrease >=15 | 9 | 10 | 5
  Heart rate >=120 and increase >=15 | 1 | 4 | 1
  Body weight decrease of >=7 percent | 7 | 8 | 4
  Body weight increase of >=7 percent | 32 | 35 | 41

2. Primary Outcome: Liver Function Tests
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) alanine aminotransferase (ALT) levels, aspartate aminotransferase levels, and bilirubin levels plus the number of participants who had ALT increases >3x ULN and ALT increases >3x ULN with concurrently increased bilirubin >1.5 ULN.
Time Frame: 4.5 years
Measure: Number; unit: participants
Arm/Group | Degarelix 240/240@40(1-3-6-9) | Degarelix 240/240@60(1-3-6-9) | Degarelix 240/240@60(1-4-7-10)
Number analyzed (Participants) | 90 | 95 | 93
participants
  Abnormal alanine aminotransferase (ALAT) | 22 | 22 | 17
  Abnormal aspartate aminotransferase | 18 | 25 | 19
  Abnormal bilirubin | 4 | 5 | 3
  ALAT >3x upper limit of normal (ULN) | 3 | 2 | 3
  ALAT >3x ULN, bilirubin >1.5x ULN | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4.5 years.
Description: Each participant's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the participant's Case Report Form.
Arm/Group | Degarelix 240/240@40(1-3-6-9) | Degarelix 240/240@60(1-3-6-9) | Degarelix 240/240@60(1-4-7-10)
Serious Adverse Events (participants affected / at risk) | 30/90 | 24/95 | 21/93
Other Adverse Events (participants affected / at risk) | 72/90 | 75/95 | 69/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240/240@40(1-3-6-9) (N=90) | Degarelix 240/240@60(1-3-6-9) (N=95) | Degarelix 240/240@60(1-4-7-10) (N=93)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Artrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mycotoxicosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Investigation (Investigations) | 1 (1) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthiritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Bladder transitional cell (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastates to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebal infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 7 (7) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (4) | 1 (1)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Arterial stenosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240/240@40(1-3-6-9) (N=90) | Degarelix 240/240@60(1-3-6-9) (N=95) | Degarelix 240/240@60(1-4-7-10) (N=93)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 7 (7) | 5 (6)
Atrial Fibrillation (Cardiac disorders) | 7 (12) | 9 (14) | 6 (6)
Cataract (Eye disorders) | 6 (8) | 1 (1) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 7 (10) | 6 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (6) | 10 (15) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4) | 6 (6) | 3 (8)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (6) | 5 (8)
Vomiting (Gastrointestinal disorders) | 3 (4) | 5 (8) | 1 (5)
Injection Site Pain (General disorders) | 24 (55) | 24 (64) | 16 (36)
Injection Site Erythema (General disorders) | 15 (29) | 14 (32) | 6 (8)
Pyrexia (General disorders) | 12 (31) | 9 (20) | 7 (22)
Fatigue (General disorders) | 10 (13) | 9 (14) | 8 (8)
Injection Site Swelling (General disorders) | 5 (12) | 10 (26) | 3 (3)
Injection Site Induration (General disorders) | 7 (7) | 4 (5) | 4 (8)
Oedema Peripheral (General disorders) | 4 (4) | 6 (6) | 4 (4)
Injection Site Nodule (General disorders) | 6 (8) | 3 (7) | 4 (6)
Injection Site Mass (General disorders) | 5 (10) | 2 (2) | 1 (1)
Injection Site Pruritus (General disorders) | 5 (6) | 2 (3) | 1 (7)
Urinary Tract Infection (General disorders) | 6 (8) | 9 (17) | 6 (6)
Nasopharyngitis (General disorders) | 5 (10) | 9 (16) | 3 (5)
Influenza (General disorders) | 4 (4) | 5 (5) | 7 (9)
Weight Increased (Investigations) | 11 (12) | 9 (10) | 7 (7)
Alanine Aminotransferase Increased (Investigations) | 6 (6) | 5 (6) | 5 (5)
Weight Decreased (Investigations) | 4 (4) | 7 (7) | 4 (4)
Aspartate Aminotransferase Increase (General disorders) | 4 (4) | 3 (4) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (13) | 7 (10) | 6 (14)
Back Pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (7) | 6 (12)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (2) | 3 (6)
Dizziness (Nervous system disorders) | 7 (9) | 9 (12) | 4 (6)
Headache (Nervous system disorders) | 5 (7) | 4 (4) | 3 (20)
Insomnia (Psychiatric disorders) | 2 (3) | 7 (7) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 5 (6) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (5) | 3 (4)
Hot Flush (Vascular disorders) | 31 (33) | 27 (29) | 32 (38)
Hypertension (Vascular disorders) | 4 (5) | 6 (6) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (3) | 5 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.